CLINICAL TRIAL: NCT05786794
Title: Hearing Healthcare Assessment in Rural Communities (HHARC)
Brief Title: Hearing Healthcare Assessment in Rural Communities
Acronym: HHARC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Bush, MD (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Matthew Bush, MD, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 65361; R33DC019602 (NIH)
Record Dates: First submitted 2023-03-14; First posted 2023-03-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Adult-Onset; Hearing Loss, Age-Related
Keywords: Patient Navigator; Adult Hearing Screening; Adult Hearing Loss
MeSH Terms: conditions — Hearing Loss; Presbycusis | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: Approximately 500 patients from 10 rural clinics will be recruited to participate in the trial. All participants will complete baseline surveys and eligible candidates will engage with a Patient Navigator who will assist them in overcoming specific barriers to obtain a diagnostic audiogram with an audiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rural Clinic Hearing Healthcare Patient Navigation Program (Experimental): This arm will involve pilot testing of the Patient Navigation Program with adults in rural primary care clinics
  Interventions: Behavioral: Patient Navigation Program for Hearing Health Care

INTERVENTIONS:
Behavioral: Patient Navigation Program for Hearing Health Care — Patients presenting for routine office visits will be invited to participate in the study and informed consent procedures and study enrollment will be conducted by a research assistant. Participants will then undergo baseline assessment. Following baseline measures, participants who screen positive for hearing loss will be contacted by the Patient Navigator (PN) to begin the intervention. The navigator will contact participants every 2 weeks to focus on addressing key aspects of Hearing Health Care (HHC): education, screening, diagnosis, and treatment. PNs will assist the patient to undergo a formal audiogram with the 12 months following enrollment. Each PN session will likely last between 10-30 minutes. Post-intervention data collection also administered by a trained interviewer, will occur following a diagnostic audiogram with an audiologist or at 12 months following enrollment.

SUMMARY:
Adult hearing loss in is the third most common chronic health condition in the United States. Adults living in rural areas face a higher risk of experiencing hearing loss, and more difficulty receiving testing and treatment than adults in urban settings. The goal of this clinical trial is to develop and test a community-based hearing healthcare patient navigation program in rural Kentucky. The main question this study aims to answer is:

-Can the number of rural adults receiving diagnostic hearing tests be increased?

DETAILED DESCRIPTION:
Investigators will pilot test the rural hearing health care patient navigation program (N=500 patients from 10 rural clinics). The program will be evaluated with the following outcome: number of participants obtaining a diagnostic audiogram within past 12 months after enrollment among rural adults

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to speak, understand, and read English.
* Patient of a participating primary care clinic

Exclusion Criteria:

-Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Receiving a Diagnostic Audiogram After Enrollment | From Enrollment to Study Completion at 12 Months
  Participants will be assisted to reduce barriers in scheduling a diagnostic audiogram within 12 months following enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Bush, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Department of Otolaryngology, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No